CLINICAL TRIAL: NCT04231240
Title: Correlation Between Hemochron and Istat in Cardiac Surgery (CHIC Study)
Acronym: CHIC
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0381
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Cardiac Event
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Adult cardiac surgery with normothermia
  Interventions: Device: Measure of ACT with IStat
- Adult cardiac surgery with hypothermia
  Interventions: Device: Measure of ACT with IStat
- Pediatric cardiac surgery with normothermia
  Interventions: Device: Measure of ACT with IStat
- Pediatric cardiac surgery with hypothermia
  Interventions: Device: Measure of ACT with IStat
- Adult cardiac surgery without cardiopulmonary bypass
  Interventions: Device: Measure of ACT with IStat

INTERVENTIONS:
Device: Measure of ACT with IStat — Measure of ACT with a point of care device named IStat

SUMMARY:
Cardiac surgery needs the use of cardiopulmonary bypass. During this time, it is necessary to prevent thrombosis with high level of heparin and to control the good efficiency with a point of care test. Investigators want to test if two different devices, Hemochron and Istat, are giving similar results.

DETAILED DESCRIPTION:
The management of the extracorporeal circulation (ECC) for cardiac surgery requires massive anticoagulation of the circuit by heparinization at 300 IU / kg of unfractionated heparin (HNF). To ensure an adequate level of safety, it is necessary to monitor the effectiveness of this dose of NHF. Several point of care monitors measuring activated coagulation time (ACT) are available on the market. Among these are the Hemochron (currently used routinely in the institution) and the IStat. These two monitors have been compared in adult cardiac surgery without deep hypothermia, but there is no comparative study in pediatric cardiac surgery.

The result of the ACT being dependent, in addition to heparinization, the platelet count, the fibrinogen level and the body temperature, it is therefore necessary to test the approval and the interchangeability between the monitors in different clinical situations .

The objective of this study is to reproduce the results published in adults and to compare these two monitors in pediatrics.

ELIGIBILITY:
Inclusion Criteria:

* adults or children
* Supported in the Department of Anesthesia - Resuscitation of the Louis Pradel Hospital (Lyon, France) for cardiac surgery with or without cardiopulmonary bypass
* Patient or Parents / Holders of parental authority informed and not opposed to participate in the study

Exclusion Criteria:

* patient with heparin-induced thrombocytopenia
* patient receiving antiplatelet therapy targeting GpIIbIIIa receptors

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with cardiac surgery with or without cardiopulmonary bypass supported in the Department of Anesthesia - Resuscitation of the Louis Pradel Hospital (Lyon, France).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Agreement of ACT measurement with Istat and Hemochron | Maximum 6 hours (time of surgery)
  Investigators will use linear regression correlation, ROC curves analysis
  Istat and Hemochron will be measured at 5 time points :
  * induction,
  * 2 minutes after heparin loading,
  * 10 minutes after the stat of cardiopulmonary bypass or after heparin,
  * 30 minutes after the start of cardiopulmonary bypass or after heparin,
  * 2 minutes after protamin
Interchangeability of ACT measurement with Istat and Hemochron | Maximum 6 hours (time of surgery)
  Investigators will use linear regression correlation, ROC curves analysis
  Istat and Hemochron will be measured at 5 time points :
  * induction,
  * 2 minutes after heparin loading,
  * 10 minutes after the stat of cardiopulmonary bypass or after heparin,
  * 30 minutes after the start of cardiopulmonary bypass or after heparin,
  * 2 minutes after protamin

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie - Réanimation de l'hôpital Louis Pradel - HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No